CLINICAL TRIAL: NCT06998043
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Nebulized Bacteriophage Treatment in Outpatient Adult Cystic Fibrosis (CF) Subjects With Chronic Pseudomonas Aeruginosa (PsA) Pulmonary Infection
Brief Title: Study With Phage for CF Subjects With Pseudomonas Lung Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BiomX Ltd (Industry)
Responsible Party: Sponsor
Organization: BiomX, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMX-04-002
Record Dates: First submitted 2025-05-10; First posted 2025-05-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pseudomonas Aeruginosa Infection; Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BX004 (Experimental): Participants will be randomized to receive standard dose of nebulized bacteriophage
  Interventions: Biological: BX004
- Placebo (Placebo Comparator): Participants will be randomized to receive nebulized placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BX004 — Bacteriophage
  Other Names: Combination of nebulized bacteriophages targeting Pseudomonas aeruginosa
  Arms: BX004
Other: Placebo — Placebo
  Other Names: Nebulized placebo
  Arms: Placebo

SUMMARY:
The goal of this Phase 2b clinical trial is to see if nebulized phage (BX004) can treat chronic Pseudomonas aeruginosa (PsA) lung infection in CF subjects. The primary goal is to see if 8 weeks of twice daily BX004 can reduce the amount of PsA in the sputum compared to placebo (on top of background CF therapy).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study to evaluate BX004 in CF subjects with chronic PsA pulmonary infection. The main purpose of the study is to evaluate whether BX004 reduces the PsA burden in the sputum of CF subjects with chronic PsA pulmonary infection. Secondary endpoints are to see how well BX004 works in improving lung function and quality of life, reducing the amount of PsA in the sputum, getting negative sputum cultures for PsA, and safety and tolerability. Clinically stable CF subjects with a confirmed diagnosis of CF and chronic PsA pulmonary infection will be enrolled. Subjects will be included in a 6-month post-dose safety follow-up. A Data Safety Monitoring Board of the CF Foundation will monitor safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Cystic fibrosis patients with chronic Pseudomonas aeruginosa pulmonary infection receiving standard of care inhaled antibiotics (cycling or continuous regimen) or no inhaled antibiotics
* Age ≥ 18 years
* FEV1 40%-80% predicted
* Clinically stable lung disease
* Willing and able to provide adequate sputum samples, using any method (spontaneously expectorated, induced, from home or clinic) at designated study visits.

Key Exclusion Criteria:

* Known hypersensitivity to bacteriophages or excipients in the formulation.
* Receipt of prior bacteriophage therapy within the 6 months prior to Screening or Day 1
* Detection of Burkholderia cenocepacia from respiratory tract within 1 year prior to Screening or from Screening culture
* Currently receiving systemic treatment for allergic bronchopulmonary aspergillosis
* Currently receiving treatment for active infection with non-tuberculous mycobacteria or prior detection of Mycobacterium abscessus in 12 months prior to Screening
* History of severe neutropenia
* History of lung transplant
* History of solid organ transplant
* Acquired or primary immunodeficiency syndrome
* Initiation or change in type of CFTR modulator less than 3 months prior to Screening
* Pregnant or breastfeeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in sputum Pseudomonas aeruginosa (PsA) burden at 8 weeks (EOT) | 8 weeks
  Change from baseline in PsA colony-forming units (CFU) per g of sputum

SECONDARY OUTCOMES:
Change in lung function at D8, D29, D43, D57 (EOT), D85, 3 months post-dose, and 6 months post-dose | from Day 8 until 6 months after last dose (end of study)
  Change from baseline in % predicted FEV1
Change from Baseline in CFQ-R respiratory domain | until 6 months after last dose of study drug
  Cystic Fibrosis Questionnaire - Revised (CFQ-R) respiratory domain: change at D29, D43, D57 (EOT), D85, 3 months post-dose, and 6 months post-dose (range 0-100; higher score=better outcome)
Change from Baseline in CFRSD-CRISS | until 6 months after last dose of study drug
  Cystic Fibrosis Respiratory Symptom Diary and Chronic Respiratory Infection Symptom Score (CFRSD-CRISS) weekly changes through D14 (daily completion), weekly changes from D21 through D85, and at 3 months post-dose, and 6 months post-dose (range 0-100; higher score=worse outcome)
Change in sputum PsA burden | until 6 months after last dose of study drug
  Change from baseline in sputum PsA CFU/g at D8, D29, D43, D85, 3 months post-dose and 6 months post-dose
Efficacy of BX004 on obtaining negative sputum cultures for PsA | until 6 months after last dose of study drug
  Proportion of subjects with negative sputum cultures for PsA, time to negative sputum cultures, durability of negative sputum cultures
Incidence of treatment-emergent adverse events [safety and tolerability] | until 6 months after last dose of study drug
  Incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — BiomX, Inc.
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Joe DiMaggio Children's Health, Hollywood, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Avanza Medical Center, Pensacola, Florida
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Medical College, Hawthorne, New York
  - Northwell Health, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Blinded clinical trial